CLINICAL TRIAL: NCT04343989
Title: A Randomized Placebo-controlled Safety and Dose-finding Study for the Use of the IL-6 Inhibitor Clazakizumab in Patients With Life-threatening COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-00392; NCT04363502 (obsolete NCT alias); NCT04659772 (obsolete NCT alias)
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — clazakizumab

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, adaptive seamless Phase II/III design (ASD). We propose the administration of an investigational drug in patients with high predicted short-term mortality secondary to COVID-19 disease. 80 patients were randomly assigned in a 1:1:1 ratio to three study arms that will receive clazakizumab at a dose of 12.5 mg, 25 mg or placebo. Interim analyses occurred every 7 days since the enrollment of the first 30 patients. Based on week 4 interim analysis the DSMB has recommendation discontinuing the low-dose 12.5 mg of clazakizumab arm. The DSMB has advised continuing enrollment in the placebo and high-dose 25mg of clazakizumab arms in a 1:1 randomization.
Who Masked: Participant, Investigator
Masking Description: This study is double-blind and therefore neither the Investigator, the subject, the Sponsor and its representatives, nor other designated study site personnel involved in running of the study will be aware of the identification of the investigational drug administered to each subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Clazakizumab 25 mg (Experimental)
  Interventions: Drug: Clazakizumab 25 mg
- Clazakizumab 12.5 mg (Experimental)
  Interventions: Drug: Clazakizumab 12.5 mg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clazakizumab 25 mg — The first dose will be administered as soon as possible after the patient is enrolled and randomized into the Clazakizumab 25 mg arm. The route of administration will be intravenous. Each dose will be administered as an infusion that is run over 30 minutes. Serum CRP will be evaluated at baseline and on days 1 and 2 following clazakizumab administration. If the CRP does not decrease by 50% within 36-48 hours after the first dose, a second dose of 25 mg clazakizumab will be given no later than day 3.
  Arms: Clazakizumab 25 mg
Drug: Clazakizumab 12.5 mg — The first dose will be administered as soon as possible after the patient is enrolled and randomized into the Clazakizumab 12.5 mg arm. The route of administration will be intravenous. Each dose will be administered as an infusion that is run over 30 minutes. Serum CRP will be evaluated at baseline and on days 1 and 2 following clazakizumab administration. If the CRP does not decrease by 50% within 36-48 hours after the first dose, a second dose of 12.5 mg clazakizumab will be given no later than day 3.
  Arms: Clazakizumab 12.5 mg
Other: Placebo — The first dose will be administered as soon as possible after the patient is enrolled and randomized into the Placebo arm. The route of administration will be intravenous. Each dose will be administered as an infusion that is run over 30 minutes. Serum CRP will be evaluated at baseline and on days 1 and 2 following clazakizumab administration. If the CRP does not decrease by 50% within 36-48 hours after the first dose, a second dose of placebo will be given no later than day 3.
  Arms: Placebo

SUMMARY:
In this study invetigators propose to administer clazakizumab to patients with life-threatening COVID-19 infection manifest by pulmonary failure and a clinical picture consistent with a cytokine storm syndrome. This is a double-blinded randomized multi-center trial designed as a phase II dose-finding three arm trial with seamless adaptive transition to a phase III efficacy trial. For phase II, patients were randomized 1:1:1 ratio to three study arms and received clazakizumab at a dose of 12.5 mg, 25 mg or placebo.

Based on interim analysis, the low dose arm was dropped and the phase III portion of the study continued to enroll patients randomized 1:1 to high dose clazakizumab or placebo.

Based on interim analysis, the remaining 10 subjects at NYU will be randomly assigned to a 1:1 ratio to two arms that will receive clazakizumab at a dose of 25 mg or placebo. The NYU site will serve as the central data management site for other centers who undertake this protocol. Other sites will enroll patients based on the two arm 1:1 randomization. 60 patients at outside sites are expected to enroll.

DETAILED DESCRIPTION:
The limited understanding of the clinical behavior of patients infected with SARS-CoV-2 (the viral organism responsible for COVID-19 disease) is evolving on a daily basis. Reports from China indicate that a subset of patients with the worst clinical outcomes may manifest cytokine storm syndrome. Hypotheses that excess cytokines may trigger a secondary hemophagocytic lymphhistiocytosis (sHLH) have been proposed. Indeed, cytokine profiles consistent with this picture were observed in Chinese patients with severe pulmonary involvement. Specifically, elevated ferritin and interleukin-6 (IL-6) were associated with fatalities among the infected patients. A role for targeted anti-inflammatory and anti-cytokine therapies in the treatment of pulmonary hyperinflammation has been proposed.

Clazakizumab is a genetically engineered humanized IgG1 monoclonal antibody (mAb) that binds with high affinity to human IL-6. This investigational agent is currently being studied as a treatment for chronic active antibody mediated rejection of renal allografts.

In this study investigators propose to administer clazakizumab to patients with life-threatening pulmonary failure secondary to COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, the patients must meet all of the following criteria:

1. At least 18 years of age
2. Confirmed COVID-19 disease (by Cobas SARS-CoV-2 real time RT-PCR using nasopharyngeal swab sample, or equivalent test available to be performed by the NYU Langone clinical laboratory). Effort will be made to have the confirmatory test result <72 hours prior to enrollment however given overall clinical demand this may not be feasible in all cases.
3. Respiratory failure manifesting as: Acute Respiratory Distress Syndrome (defined by a P/F ratio of <200), OR SpO2 < 90% on 4L (actual or expected given higher O2 requirement) OR increasing O2 requirements over 24 hours, PLUS 2 or more of the following predictors for severe disease:

   CRP > 35 mg/L Ferritin > 500 ng/mL D-dimer > 1000 mg/mL Neutrophil-Lymphocyte Ratio > 4 LDH > 200 U/L Increase in troponin in patient w/out known cardiac disease
4. Has a consent designee willing to provide informed consent on behalf of the patient (this assumes that a mechanically ventilated patients lacks capacity to consent on his/her own behalf. Should it be deemed that the patient has capacity to consent, consent may be obtained from the patient.)
5. Women of childbearing potential must be willing and able to use at least one highly effective contraceptive method for a period of 5 months following the study drug administration. In the context of this study, an effective method is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly such as:

   1. combined (estrogen and progestogen containing) hormonal contraception combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, or transdermal)
   2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
   3. intrauterine device (IUD)
   4. intrauterine hormone-releasing system (IUS)
   5. vasectomized partner
   6. bilateral tubal occlusion
   7. true abstinence. when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence, such as calendar, ovulation, symptothermal, postovulation methods, and withdrawal are not acceptable methods of contraception.
6. Men must be willing to use a double-barrier contraception from enrollment until at 5 months after the last dose of study drug, if not abstinent.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Evidence of irreversible injury deemed non-survivable even if the pulmonary failure recovers (for example severe anoxic brain injury)
2. Known active inflammatory bowel disease
3. Known active, untreated diverticulitis
4. Known untreated bacteremia
5. Pregnancy. (The protocol will exclude pregnant subjects given the lack of overall data on use of clazakizumab in pregnancy however the study team would consider a protocol revision should more than 3 potential pregnant study subjects be excluded on this basis).
6. Known hypersensitivity to the clazakizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Lonze, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - New York University School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Upon reasonable request by an investigator who proposes to use the data.

REFERENCES:
- [Derived] Lonze BE, Spiegler P, Wesson RN, Alachkar N, Petkova E, Weldon EP, Dieter RA, Li Y, Quinn M, Mattoo A, Soomro I, Cohen SM, Leung S, Deterville CL, Landrum BM, Ali MI, Cohen DJ, Singer AL, Sen A, Chong E, Hochman JS, Troxel AB, Montgomery RA. A Randomized Double-Blinded Placebo Controlled Trial of Clazakizumab for the Treatment of COVID-19 Pneumonia With Hyperinflammation. Crit Care Med. 2022 Sep 1;50(9):1348-1359. doi: 10.1097/CCM.0000000000005591. Epub 2022 May 17. PMID 35583232

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Started | 78 | 26 | 74
Completed | 78 | 26 | 74
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo | Total
Number analyzed (Participants) | 78 | 26 | 74 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (11.1) | 65.7 (8.3) | 59.8 (13.1) | 62.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 10 | 20 | 55
  Male | 53 | 16 | 54 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 8 | 24 | 49
  Not Hispanic or Latino | 61 | 18 | 50 | 129
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 2 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 4 | 12 | 32
  White | 25 | 14 | 27 | 66
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 30 | 6 | 26 | 62
Region of Enrollment [Number; unit: participants]
  United States | 78 | 26 | 74 | 178

OUTCOME MEASURES:

1. Primary Outcome: Ventilator Free Survival
Description: Ventilator Free Survival is defined as the total number of patients who were alive and ventilator free at 28 days.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Number analyzed (Participants) | 78 | 26 | 74
Participants | 58 | 19 | 44

2. Primary Outcome: Number of Serious Adverse Events Associated With High and Low Dose of Clazakizumab
Time Frame: 60 days
Measure: Number; unit: Serious Adverse Events
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Number analyzed (Participants) | 78 | 26 | 74
Serious Adverse Events | 46 | 6 | 51

3. Secondary Outcome: Overall Patient Survival
Description: Overall Patient Survival is defined as the total number of patients per group who were alive at 28 days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Number analyzed (Participants) | 78 | 26 | 74
Participants | 60 | 20 | 54

4. Secondary Outcome: Overall Patient Survival
Description: Overall patient survival is defined as total number of patients per group who were alive at 60 days.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Number analyzed (Participants) | 78 | 26 | 74
Participants | 56 | 20 | 46

5. Secondary Outcome: Number of Participants With Change in Clinical Status
Description: Change in clinical status defined by an improvement in status by at least 2 score points on WHO 11-point ordinal scale, where 0 = uninfected; no viral RNA detected, 1 = asymptomatic; viral RNA detected, 2 = symptomatic; independent, 3 = symptomatic; assistance needed, 4 = hospitalized; no oxygen therapy, 5 = hospitalized; oxygen by mask or nasal prongs, 6 = hospitalized; oxygen by NIV or high flow, 7 = intubation and mechanical ventilation, pO2/FiO2 >/= 150 or SpO2/FiO2 >/= 200, 8 = mechanical ventilation pO2/FiO2 < 150 (SpO2/FiO2 < 200) or vasopressors, 9 = mechanical ventilation pO2/FiO2 < 150 and vasopressors, dialysis, or ECMO, and 10 = Dead
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Number analyzed (Participants) | 78 | 26 | 74
Participants | 50 | 15 | 37

6. Secondary Outcome: Number of Participants With a Change in Clinical Status
Description: as for outcome 5
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Number analyzed (Participants) | 78 | 26 | 74
Participants | 54 | 17 | 40

7. Secondary Outcome: Number of Clazakizumab-expected Adverse Events
Time Frame: 60 days
Measure: Number; unit: Adverse Events
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
Number analyzed (Participants) | 78 | 26 | 74
Adverse Events | 7 | 3 | 12

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Clazakizumab 25 mg | Clazakizumab 12.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 22/78 | 6/26 | 28/74
Serious Adverse Events (participants affected / at risk) | 24/78 | 6/26 | 33/74
Other Adverse Events (participants affected / at risk) | 76/78 | 24/26 | 72/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clazakizumab 25 mg (N=78) | Clazakizumab 12.5 mg (N=26) | Placebo (N=74)
acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0
adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
alanine aminotransferase increased (Hepatobiliary disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
aspartate aminotransferase increased (Hepatobiliary disorders) | 0 | 0 | 1
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
bacteremia (Infections and infestations) | 1 | 0 | 0
bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
cardiac arrest (Cardiac disorders) | 14 | 6 | 19
gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
heart failure (Cardiac disorders) | 0 | 0 | 1
hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
hypotension (General disorders) | 1 | 0 | 3
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
infections (Infections and infestations) | 0 | 0 | 1
intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1
lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
lymphocyte count increased (Blood and lymphatic system disorders) | 1 | 0 | 0
multi-organ failure (General disorders) | 2 | 0 | 0
muscle weakness (Nervous system disorders) | 1 | 0 | 0
platelet count decreased (Blood and lymphatic system disorders) | 1 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 7
sepsis (Infections and infestations) | 2 | 0 | 1
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
urinary tract infection (Infections and infestations) | 1 | 0 | 0
visceral arterial ischemia (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clazakizumab 25 mg (N=78) | Clazakizumab 12.5 mg (N=26) | Placebo (N=74)
abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
acidosis (Metabolism and nutrition disorders) | 4 | 2 | 5
alanine aminotransferase increased (Hepatobiliary disorders) | 18 | 4 | 21
alkaline phosphatase increased (Hepatobiliary disorders) | 4 | 0 | 6
alopecia (General disorders) | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 17 | 11 | 32
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 0 | 1
aspartate minotransferase increased (Hepatobiliary disorders) | 10 | 0 | 11
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 12
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bacteremia (Infections and infestations) | 4 | 1 | 6
blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 | 0 | 1
blood bilirubin increased (Hepatobiliary disorders) | 4 | 0 | 4
Blurred vision (Nervous system disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 2
bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
bronchopulmonary hemorrahge (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 2 | 1
cardiac troponin increased (Cardiac disorders) | 2 | 0 | 0
chest pain-cardiac (Cardiac disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
cognitive disturbance (Nervous system disorders) | 0 | 0 | 1
Confusion (Nervous system disorders) | 1 | 0 | 0
creatinine increased (Renal and urinary disorders) | 14 | 9 | 25
cystitis (Renal and urinary disorders) | 0 | 0 | 1
cytomegalovirus infection (Infections and infestations) | 0 | 0 | 2
dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
delirium (Nervous system disorders) | 2 | 1 | 3
depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 2
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
dysphagia (Nervous system disorders) | 0 | 0 | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
encephalopathy (Nervous system disorders) | 1 | 1 | 0
eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
epistaxis (General disorders) | 1 | 0 | 2
fall (General disorders) | 3 | 1 | 1
fever (General disorders) | 24 | 16 | 59
fibrinogen decreased (Blood and lymphatic system disorders) | 1 | 0 | 0
fungemia (Infections and infestations) | 1 | 0 | 0
gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1
hematoma (General disorders) | 3 | 0 | 2
hematuria (Renal and urinary disorders) | 1 | 0 | 1
hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 1
hepatobiliary disoders, other (Hepatobiliary disorders) | 0 | 0 | 1
herpes simplex reactivation (Infections and infestations) | 0 | 1 | 0
hyperglycemia (Endocrine disorders) | 2 | 0 | 1
hyperkalemia (Metabolism and nutrition disorders) | 8 | 2 | 12
hyperlipidemia (Metabolism and nutrition disorders) | 2 | 0 | 4
hypermagnesemia (Metabolism and nutrition disorders) | 5 | 0 | 4
hypernatremia (Metabolism and nutrition disorders) | 5 | 1 | 3
hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 1
hypertension (General disorders) | 1 | 0 | 0
hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 0 | 6
hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 5
hyponatremia (Metabolism and nutrition disorders) | 5 | 0 | 6
hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0 | 3
hypotension (General disorders) | 24 | 16 | 42
hypothermia (General disorders) | 3 | 0 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 29
ileus (Gastrointestinal disorders) | 1 | 0 | 1
inr increased (Blood and lymphatic system disorders) | 2 | 0 | 0
intracranial hemorrhage (Nervous system disorders) | 1 | 1 | 0
lethargy (Nervous system disorders) | 0 | 0 | 1
lower gastrointestinal hemorrahge (Gastrointestinal disorders) | 2 | 0 | 0
lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 9
lymphocyte count decreased (Blood and lymphatic system disorders) | 10 | 0 | 8
maculopapular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 | 0 | 1
muscle weakness (Nervous system disorders) | 0 | 0 | 3
nasal congestion (General disorders) | 1 | 0 | 1
neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 0 | 0
non-cardiac chest pain (General disorders) | 0 | 0 | 1
oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 8
paresthesia (Nervous system disorders) | 0 | 0 | 1
pericardial effusion (Cardiac disorders) | 1 | 0 | 0
peripheral ischemia (Vascular disorders) | 2 | 0 | 3
peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Platelet Count Decreased (Blood and lymphatic system disorders) | 12 | 1 | 5
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 15
presyncope (Nervous system disorders) | 1 | 0 | 0
proteinuria (Renal and urinary disorders) | 0 | 0 | 1
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
renal calculi (Renal and urinary disorders) | 0 | 1 | 0
retroperitoneal hemhorrahge (General disorders) | 1 | 0 | 0
right ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
seizure (Nervous system disorders) | 2 | 0 | 2
sepsis (Infections and infestations) | 2 | 0 | 0
sinus bradycardia (Cardiac disorders) | 2 | 1 | 2
sinus tachycardia (Cardiac disorders) | 4 | 1 | 10
skin & subcutaneous tissue disorders (Infections and infestations) | 1 | 0 | 0
skin infection (Infections and infestations) | 1 | 0 | 0
skin ulceration (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
soft tissue infection (Infections and infestations) | 0 | 0 | 1
soft tissue necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
somnolence (Nervous system disorders) | 1 | 1 | 1
sore throat (Gastrointestinal disorders) | 1 | 0 | 0
stroke (Nervous system disorders) | 2 | 0 | 5
subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
tachycardia (Cardiac disorders) | 2 | 0 | 1
tachypnic (Cardiac disorders) | 0 | 0 | 1
thromboembolic event (Blood and lymphatic system disorders) | 3 | 3 | 6
thrush (Gastrointestinal disorders) | 0 | 0 | 1
tracheal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
triglycerides increased (Metabolism and nutrition disorders) | 1 | 0 | 0
upper gastrointestinal hemorrahge (Gastrointestinal disorders) | 4 | 0 | 1
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 12
urinary frequency (Renal and urinary disorders) | 0 | 0 | 1
urinary retention (Renal and urinary disorders) | 2 | 2 | 1
urinary tract infection (Infections and infestations) | 2 | 0 | 10
ventricular tachycardia (Cardiac disorders) | 3 | 0 | 0
vomiting (Gastrointestinal disorders) | 1 | 0 | 1
weight loss (Metabolism and nutrition disorders) | 0 | 0 | 1
multi-organ failure (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04343989/Prot_SAP_000.pdf